CLINICAL TRIAL: NCT04739267
Title: The Acute Coronary Syndrome Accelerated CardioFlux TM Magnetocardiography-based Early Disposition Study
Brief Title: Acute Coronary Syndrome CardioFlux TM Study (ACCMED)
Acronym: MAGNETO
Status: Completed | Type: Observational
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1000-2
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Acute Myocardial Injuries
Keywords: Ischemia; Cardiovascular Disease; MCG; CardioFlux
MeSH Terms: conditions — Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: CardioFlux — Not an intervention

SUMMARY:
Approximately 16.5 million people suffer from coronary artery disease (CAD) and about 10 million present each year to emergency departments with symptoms like chest pain and shortness of breath, commonly suggestive of acute coronary syndrome (ACS). To clinically assess ACS risk in these patients, there are typically 2-6 hours of emergency room evaluation, followed by 6-42 hours of an observation period prior to discharge. The clinical pathway includes: 1) 1-3 ECG's; 2) serial troponins (1 and 3 hours vs 1 and 6 hours); and 3) other pertinent diagnostic information, including but not limited to echocardiography, stress testing and/or CT Angiography. Patients who are evaluated, have presented with a low risk for ACS, and maintain negative diagnostic results can potentially be discharged within 6 hours. However, 20%-40% of patients who fall into indeterminate diagnostic categories will require longer observation periods or admission of 12-48 hours which result in the use of expensive imaging and provocative testing, such as stress testing. The purpose of ACCMED is to measure the efficacy of Magnetocardiography (MCG) as a diagnostic tool to rule-in/rule-out myocardial ischemia in patients with suspicion of an acute coronary syndrome who have a HEART Score > 2 and to allow safe and timely disposition of the patient to an appropriate level of care.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of enrollment.
2. Patient presenting acutely with signs and symptoms suggestive of ACS.
3. Informed Consent Form signed by subject or LAR.
4. HEART Score of >2.
5. Patient consented within 4 hours of the beginning of the clinical assessment (exclusive of any screening examination) for suspected ACS by an appropriately credentialed clinician.

Exclusion Criteria:

1. < 18 years of age.
2. STEMI.
3. Unable to fit into device.
4. Non-ambulatory patients.
5. Positive response on MCG metal checklist.
6. Deemed hemodynamically unstable by treating physician, regardless of cause.
7. Unable to lie supine for up to 5 minutes.
8. Poor candidate for follow-up (e.g., no access to phone).
9. Prisoners.
10. Repeat participants.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the ED with symptoms of potential ACS and fitting the eligibility/exclusion criteria will be approached for accrual
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
To prove that MCG can accurately diagnose myocardial ischemia | 1 year
  Demonstrate the following:
  1. MCG has a clinically acceptable sensitivity and specificity for the detection of myocardial ischemia. This will be compared to the Gold Standard of index revascularization, ≥70% stenosis in any coronary artery as determined by invasive coronary angiography, or 30-day MACE.
  2. MCG is non-inferior to noninvasive downstream testing (DS) for the identification of patients with myocardial ischemia.
  3. MCG is non-inferior to noninvasive downstream testing (DS) for appropriate referral of patients to invasive coronary angiography with decision to refer the patient to the coronary catheterization laboratory as the Gold Standard.

SECONDARY OUTCOMES:
To demonstrate that MCG provides value to the traditional HEART score for risk stratification of patients with suspected ACS. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Mace, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Genetesis Facility, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Yang G, Yao Y, Du Y, Huang J. Cardiac troponin had limited diagnostic value for acute myocardial infarction in renal insufficiency: a meta-analysis. Biomark Med. 2020 Apr;14(6):481-493. doi: 10.2217/bmm-2019-0339. Epub 2020 Apr 9. PMID 32270694
- [Background] Chiang CH, Chiang CH, Lee GH, Gi WT, Wu YK, Huang SS, Yeo YH, Giannitsis E, Lee CC. Safety and efficacy of the European Society of Cardiology 0/1-hour algorithm for diagnosis of myocardial infarction: systematic review and meta-analysis. Heart. 2020 Jul;106(13):985-991. doi: 10.1136/heartjnl-2019-316343. Epub 2020 Apr 3. PMID 32245882
- [Background] Lee CC, Huang SS, Yeo YH, Hou YT, Park JY, Inoue K, Hsu WT. High-sensitivity-cardiac troponin for accelerated diagnosis of acute myocardial infarction: A systematic review and meta-analysis. Am J Emerg Med. 2020 Jul;38(7):1402-1407. doi: 10.1016/j.ajem.2019.11.035. Epub 2019 Dec 28. PMID 31932131
- [Background] Madsen TE, Stewart M, Smyres C, Beal A, Hamilton D, Vlasic K, Oates A. Significance of an Indeterminate Troponin I in Patients Evaluated for Chest Pain in an Emergency Department Observation Unit. Crit Pathw Cardiol. 2015 Dec;14(4):146-9. doi: 10.1097/HPC.0000000000000054. PMID 26569654
- [Background] Madsen T, Perkins R, Holt B, Carlson M, Steenblik J, Bossart P, Hartsell S. Emergency Department Observation Unit Utilization Among Older Patients With Chest Pain. Crit Pathw Cardiol. 2019 Mar;18(1):19-22. doi: 10.1097/HPC.0000000000000166. PMID 30747761